CLINICAL TRIAL: NCT04876417
Title: Transcranial Direct Current Stimulation (tDCS) for the Treatment of Fatigue in Post-COVID-19 Patients
Brief Title: Transcranial Direct Current Stimulation (tDCS) for Post COVID-19 Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202009381
Record Dates: First submitted 2021-03-15; First posted 2021-05-06 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Post Covid-19 Patients
Keywords: Covid-19; Fatigue
MeSH Terms: conditions — COVID-19; Fatigue | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- tDCS and fatigue (Active Comparator): This group will receive the active form of tDCS.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham and fatigue (Sham Comparator): This group will receive the sham form of tDCS.
  Interventions: Device: Sham Transcranial Direct Current Stimulation
- tDCS and non-fatigue (Active Comparator): This group will receive the active form of tDCS.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham and non-fatigue (Sham Comparator): This group will receive the sham form of tDCS.
  Interventions: Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial Direct Current Stimulation is a form of non-invasive brain stimulation. It uses small electrodes to deliver small amounts of current to specific areas of the brain to either increase or decrease excitability.
  Other Names: tDCS
  Arms: tDCS and fatigue; tDCS and non-fatigue
Device: Sham Transcranial Direct Current Stimulation — Transcranial Direct Current Stimulation is a form of non-invasive brain stimulation. It uses small electrodes to deliver small amounts of current to specific areas of the brain to either increase or decrease excitability.
  Other Names: tDCS
  Arms: Sham and fatigue; Sham and non-fatigue

SUMMARY:
The objective of this study is to investigate the short- and long-term effects of multiple sessions of 4 mA M1 tDCS on fatigue and brain activity in recovered COVID-19 patients using established measures of perception of fatigue, performance fatigability, and cerebral glucose uptake. Our central hypothesis is that tDCS will improve fatigue short- and long-term, and thus will improve quality of life (QOL) in recovered COVID-19 patients and that these changes will be associated with alterations in brain activity.

DETAILED DESCRIPTION:
For survivors of severe COVID-19, overcoming the virus is just the beginning of an uncharted recovery path. As the number of confirmed COVID-19 cases exceeds 27 million globally and 6 million in the US, the number of patients who experience persistent symptoms during recovery is rapidly growing. In COVID-19 patients, common acute symptoms include cough, fever, dyspnea, musculoskeletal symptoms (myalgia, joint pain, fatigue), gastrointestinal symptoms, and anosmia/dysgeusia . Clinicians and researchers have focused on the acute phase of COVID-19, but continued monitoring and treating of persistent symptoms is urgently needed. Recent studies assessed persistent symptoms in patients who were discharged from the hospital after recovering from COVID-19. None of the patients had a fever or any of the other signs or symptoms associated with acute illness. Nevertheless, decreased quality of life was observed in 44.1% and fatigue was reported by 53.1% and 71% of patients. Furthermore, persistent fatigue following COVID-19 infection is common and independent of severity of initial infection (hospitalized and non-hospitalized patients). In addition to the characteristic laboratory findings and lung computed tomography (CT) abnormalities, it has been recently reported that patients with COVID-19 also have neurological manifestations. Wu et al. [2020] found that viral infections have detrimental impacts on neurological functions and can even cause severe neurological damage. Their study showed that coronaviruses (CoV), especially severe acute respiratory syndrome CoV 2 (SARS-CoV-2), exhibited neurotropic properties and may cause neurological diseases with severe fatigue symptoms. Another recent case report has also indicated reduced glucose uptake ([18F]flurodeoxyglucose (FDG); measured with positron emission tomography (PET)) in diverse brain areas [9], which may contribute to these neurological manifestations. Therefore, there is a critical need to develop inexpensive, effective, and rapid treatments for the persistent fatigue experienced by recovered COVID-19 patients. Without such treatments, these patients will continue to experience fatiguing symptoms that significantly reduce their quality of life. One possible treatment modality is transcranial direct current stimulation (tDCS) [10]. tDCS uses weak currents applied to the scalp to alter the excitability of cortical neurons by changing their spontaneous firing rate. It also has a favorable safety profile and only transient adverse side effects. Studies in patients with neurological disorders have shown that tDCS over the primary motor and/or sensory cortex (M1/S1) consistently and significantly improves fatigue. M1 tDCS represents an easy, cost-effective candidate for treating persistent fatigue in recovered COVID-19 patients.

ELIGIBILITY:
Only those that are discharged from the UIHC COVID-19 inpatient clinic and/or that meet the CDC guidelines for discontinuing home isolation (i.e., fever free for at least 24 hours, all symptoms improved after 10 days) will initially be considered as long as they meet the rest of the following criteria:

Inclusion criteria

1. 18-80 yrs.
2. Meet CDC guidelines (https://www.cdc.gov/coronavirus/2019-ncov/hcp/duration-isolation.html) for discontinuation of home isolation
3. Meet the criteria for fatigue, based on the Chalder Fatigue Scale CFQ-11 case definition of fatigue
4. Healthy enough to complete the protocol based, on information obtained from a clinical exam and past medical history, such as cardiovascular disease.
5. Comprehension of the protocol, as indicated by an ability to respond to questions about the study after reading the consent form.
6. Able to use and be contacted by telephone
7. Able to speak, read, and understand English, and complete questionnaires in English

Exclusion criteria

1. Medical diagnosis or condition that is considered to be an absolute or relative contraindication to participating in exercise training, such as major renal, pulmonary, hepatic, cardiac, gastrointestinal, HIV, cancer (other than treated basal cell cancer), or neurological disorders
2. History/presence of secondary conditions such as seizure disorders (or on medications known to lower seizure threshold), hydrocephalus, diabetes mellitus, or claustrophobia
3. Alcohol dependence or abuse (>2 drinks/day), or present history of drug abuse (last six months)
4. History of significant traumatic brain injury or hydrocephalus
5. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Health and Human Physiology, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham and Fatigue; Sham and Non-fatigue: This group will receive the sham form of tDCS.
  Transcranial Direct Current Stimulation: Transcranial Direct Current Stimulation is a form of non-invasive brain stimulation. It uses small electrodes to deliver small amounts of current to specific areas of the brain to either increase or decrease excitability.
Period: Overall Study
Arm/Group | tDCS and Fatigue | Sham and Fatigue | tDCS and Non-fatigue | Sham and Non-fatigue
Started | 27 | 27 | 10 | 10
Completed | 22 | 19 | 10 | 10
Not Completed | 5 | 8 | 0 | 0
Not completed — Lost to Follow-up | 5 | 8 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Post-COVID fatigue
Groups:
- Sham and Fatigue; Sham and Non-fatigue: This group will receive the sham form of tDCS.
  Sham Transcranial Direct Current Stimulation
- Total: Total of all reporting groups
Arm/Group | tDCS and Fatigue | Sham and Fatigue | tDCS and Non-fatigue | Sham and Non-fatigue | Total
Number analyzed (Participants) | 22 | 19 | 10 | 10 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 19 | 10 | 10 | 61
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.23 (11.71) | 36.74 (14.37) | 30.13 (10.02) | 30.13 (10.02) | 34.30 (14.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 6 | 7 | 43
  Male | 6 | 5 | 4 | 3 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 2 | 5
  Not Hispanic or Latino | 21 | 17 | 10 | 8 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 1 | 3
  White | 17 | 17 | 9 | 6 | 49
  More than one race | 2 | 1 | 0 | 1 | 4
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 19 | 10 | 10 | 61

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Assessment Scale (FAS)
Description: Fatigue Questionnaire (1 to 5-point scale x 10 questions for a total score range of 0 to 50) where a low value indicates less fatigued (better outcome) and a high value indicates more fatigued (worse outcome)
Time Frame: through study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: Total score (1 to 5 point scale)
Groups:
- tDCS and Non-fatigue: This group will receive the active form of tDCS. Transcranial Direct Current Stimulation: Transcranial Direct Current Stimulation is a form of non-invasive brain stimulation. It uses small electrodes to deliver small amounts of current to specific areas of the brain to either increase or decrease excitability.
Arm/Group | tDCS and Fatigue | Sham and Fatigue | tDCS and Non-fatigue | Sham and Non-fatigue
Number analyzed (Participants) | 22 | 19 | 10 | 10
Total score (1 to 5 point scale) | 31.32 (8.41) | 28.42 (6.41) | 14.90 (3.63) | 15.3 (4.57)

2. Primary Outcome: Fatigue Severity Scale (FSS)
Description: Fatigue Questionnaire (1 to 7 point scale x 9 questions for a total score range of 0 to 63) with a low value indicating less severe fatigue (better outcome) and a high value indicating more severe fatigue (worse outcome)
Time Frame: through study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: Total score (1-7 point scale)
Arm/Group | tDCS and Fatigue | Sham and Fatigue | tDCS and Non-fatigue | Sham and Non-fatigue
Number analyzed (Participants) | 22 | 19 | 10 | 10
Total score (1-7 point scale) | 5.08 (1.60) | 4.73 (1.14) | 2.13 (0.61) | 1.98 (0.55)

3. Primary Outcome: 6-minute Walk Test
Description: Distance in meters will be measured in six minutes
Time Frame: through study completion, an average of 8 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | tDCS and Fatigue | Sham and Fatigue | tDCS and Non-fatigue | Sham and Non-fatigue
Number analyzed (Participants) | 22 | 19 | 10 | 10
meters | 435.4 (70.47) | 460.69 (58.67) | 489.01 (68.11) | 451.38 (65.86)

ADVERSE EVENTS:
Time Frame: 1 month
Description: Does not differ
Groups:
- tDCs and Non-fatigued: This group will receive the active form of tDCS.
  Transcranial Direct Current Stimulation: Transcranial Direct Current Stimulation is a form of non-invasive brain stimulation. It uses small electrodes to deliver small amounts of current to specific areas of the brain to either increase or decrease excitability.
- Sham and Non-fatigued: This group will receive the sham form of tDCS.
  Transcranial Direct Current Stimulation: Transcranial Direct Current Stimulation is a form of non-invasive brain stimulation. It uses small electrodes to deliver small amounts of current to specific areas of the brain to either increase or decrease excitability.
Arm/Group | tDCS and Fatigue | Sham and Fatigue | tDCs and Non-fatigued | Sham and Non-fatigued
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT04876417/Prot_SAP_000.pdf